CLINICAL TRIAL: NCT05742880
Title: Effect of Face Masks on Pulmonary Function in Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Lukasz Antoniewicz, MD, PhD, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1163/2022
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: COPD; Walking, Difficulty
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Mobility Limitation | interventions — Blood Gas Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Without Facemask (Sham Comparator): Wearing no mask.
  Interventions: Diagnostic Test: 6 Minute Walking Test; Diagnostic Test: Blood gas analysis; Procedure: Wearing no Mask
- Wearing a Facemask (Active Comparator): Wearing a surgical facemask
  Interventions: Diagnostic Test: 6 Minute Walking Test; Diagnostic Test: Blood gas analysis; Procedure: Wearing a Surgical Facemask
- Wearing a FFP2-Mask (Active Comparator): Wearing a FFP2- Mask
  Interventions: Diagnostic Test: 6 Minute Walking Test; Diagnostic Test: Blood gas analysis; Procedure: Wearing a FFP2- Facemask

INTERVENTIONS:
Diagnostic Test: 6 Minute Walking Test — 6 Minute walking test
Diagnostic Test: Blood gas analysis — Blood gas analyisis
Procedure: Wearing a Surgical Facemask — Wearing a Surgical Facemask
  Arms: Wearing a Facemask
Procedure: Wearing a FFP2- Facemask — Wearing a FFP2- Facemask
  Arms: Wearing a FFP2-Mask
Procedure: Wearing no Mask — Wearing no Mask
  Arms: Without Facemask

SUMMARY:
Given the heightened vulnerability of COPD patients to severe illness upon SARS-CoV-2 infection, precautions like mask-wearing are deemed crucial. Yet, mask-wearing can exacerbate breathlessness and discomfort in this demographic. This study aims to assess the effects of wearing a face mask during 6-Minute-Walking-Tests (6-MWT) among COPD patients.

DETAILED DESCRIPTION:
In this detailed study, we aim to explore the impact of wearing face masks on COPD patients during 6-Minute-Walking-Tests (6MWT). COPD, commonly observed among smokers and former smokers, poses heightened mortality risks upon SARS-CoV-2 infection. Consequently, face masks are often recommended for preventive measures. However, breathlessness remains a predominant symptom in this patient cohort. Moreover, there is a dearth of data concerning blood oxygenation levels while wearing various types of face masks.

The study will involve COPD patients who will undergo three 6MWTs: one without a mask, one with a simple face mask, and one with a FFP2 mask. Prior to each 6MWT, comprehensive pulmonary function tests including spirometry, body plethysmography, and CO-diffusion capacity measurement will be conducted. Additionally, capillary blood gas analysis will be performed both before the 6MWT and after each test session.

ELIGIBILITY:
Inclusion Criteria:

* COPD Diagnosis
* Vaccinated against SARS-CoV 2

Exclusion Criteria:

* Known cardial insufficency
* Long term oxgenation therapy
* immobility
* BMI >35
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Walking distance | 6 minutes
  Walking distance in meters during a 6 minute walking test

SECONDARY OUTCOMES:
Blood oxygenation | 6 minutes
  Blood oxygenation
Heart rate | 6 minutes
  Heart rate in bpm
pO2 | 6 minutes
  pO2

CONTACTS AND LOCATIONS:
Overall Officials: Marco Idzko, Prof., Study Chair — Medical University of Vienna; Lukasz Antoniewicz, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Dept. of Internal Medicine II, Div. of Pulmonology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No